CLINICAL TRIAL: NCT02086747
Title: The Management of Chronic Pain With Acetaminophen Four Times a Day
Brief Title: Acetaminophen for Chronic Pain in Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Asist.Prof, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/33
Record Dates: First submitted 2014-02-07; First posted 2014-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
Keywords: Abdominal Hysterectomy, Acetaminophen, chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Active Comparator): Postoperative 72 hours acetaminophen 1 g iv 4 times a day for 72 hours iv
  Interventions: Drug: Acetaminophen
- isotonic (Placebo Comparator): 1 g intravenous %0.9 NaCl four times Daily for 72 hours
  Interventions: Drug: Isotonic

INTERVENTIONS:
Drug: Acetaminophen — 100 ml iv, 4 times a day for 72 hours
  Other Names: Parol
  Arms: Acetaminophen
Drug: Isotonic — 100 ml iv, 4 times a day for 72 hours
  Arms: isotonic

SUMMARY:
The investigators hypothesized that 1 mg of acetaminophen 4 times per day for 3 days prevent chronic pain in hysterectomy patients.

DETAILED DESCRIPTION:
The most appropriate expression of the pain is "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage" (IASP,2008) (1). When pain lasts longer than 3 months or beyond the time when an acute injury would be expected to have healed, the patient's presentation becomes more complex, often, not surprisingly, with more psychological features. These include complaints of poor or non-refreshing sleep, tiredness, depression and poor concentration. Pain at this stage is often said to be "chronic" (2). Chronic pain is not only a common problem but also a significant and increasing public health burden in virtually all developed countries (3). Hysterectomy is one of the most common surgical procedures in women. Recent studies have recognized that there is a 20-40% incidence of chronic post-surgical pain after hysterectomy surgery (4)(5)(6). Effective pain management is an important component of postsurgical care. Many patients, however, continue to experience inadequate pain relief (7) Despite all analgesic strategies, in the postoperative periods 80% of patients still suffer from moderate to severe pain (8).

The ideal analgesic has some properties like rapid and effective pain relief, minimal adverse effects, and minimal impact on major organ systems or no interaction with other pharmacologic agents. Opioids are still good choice for postoperative pain but has dose dependent adverse effects and negative postoperative outcomes (9)(10). Nonopioid analgesics are commonly used alone or as adjuncts to opioid-based analgesia to treat moderate to severe pain. Perioperative administration of acetaminophen with nonsteroidal antiinflammatory drugs (NSAIDs) has been advocated to provide "multimodal" or "balanced" analgesia that decreases opioid dose requirements and may reduce associated adverse events while reducing postsurgical pain intensity ( 9)(11). Acetaminophen is superior to the other analgesics because of safety and analgesic profile. At the same time it has less contraindications and drug interactions with the others. Acetaminophen act by selectively inhibiting the release of prostaglandins within the central nervous system as well as having some peripheral analgesic effect (12). Rarely overdose use can induce hepatoxicity (13).

While providing fast and significant pain relief as well as a significant morphine-sparing effect,(14) (15). it is not associated with the increased incidence of nausea, vomiting, and respiratory depression observed with opioids or the deleterious gastrointestinal, hematologic, and renal effects associated with NSAIDs and cyclooxygenase (COX)-2 inhibitors (16).

Several international guidelines (EULAR, ACR) and influential reviews recommend the use of paracetamol as the first-line analgesic of choice for the management of chronic pain, as it provides cost-effective analgesia without the risks associated with NSAID use, particularly in the elderly. Based on currently available data, the use of alternative analgesics, such as tramadol and opioids, either alone or in combination with paracetamol, is warranted in those patients whose pain does not respond to nonnarcotic analgesics. While these recommendations are based on a vast amount of clinical data, they do not account for individual patient responses (17).

Paracetamol is rapidly absorbed from immediaterelease formulations, with maximum concentrations in plasma typically occurring between 0.25 and 2.0 hours, and an onset of action within about 30 minutes (18). Because the terminal elimination phase half-life of paracetamol in plasma is short, in the region of 1.9-2.5 hours after a therapeutic dose,(19) the recommended time between doses is 4-6 hours, resulting in a 4-times daily dosing schedule.

The investigators hypothesised that postoperative treatment with paracetamol with repeated doses of 1 g in comparison of placebo in hysterectomy patients with moderate or severe pain would decrease analgesics consumption perioperatively and the incidence of chronic pain associated with abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years old scheduled for hysterectomy
* Horizontal or vertical abdominal skin incision
* Ability to operate a patient-controlled analgesia (PCA) device
* Written informed consent.

Exclusion Criteria:

* ASA Physical Status I-II, emergency or urgent procedure
* Pre-existing chronic pain (at any site) requiring opioid analgesia
* History of significant Axis I psychiatric disease (major depressive disorder, bipolar disorder, schizophrenia, etc.)
* Significant hepatic (ALT or AST > 2 times normal) or renal (serum creatinine > 2 mg/dl) impairment; allergy to acetaminophen
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Acetaminophen prevents postoperative chronic pain in hysterectomy patients | postoperative 3.months

SECONDARY OUTCOMES:
Postoperative pain | postoperative 0h, 1h, 4h, 8h, 12h, 16h, 20h, 24hours.
  After hysterectomy operations, postoperative pain is really high. Assesment and intervention to pain in postoperative period is important. We use narcotics in PCA and diclofenac in both groups also acetaminophen 1 g 4 times per day for 72 hours in one group.

OTHER OUTCOMES:
Postoperative complications and ramsey sedation scores | Postoperative 24 hours
  Postoperative complications and ramsey sedation scales are assessed in postoperative 0h, 1h, 4h, 8h, 12h, 16h, 20h, 24hours.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Koyuncu, Asist.Prof, Study Chair — Mustafa Kemal University
Locations (1):
- Mustafa Kemal University Medicine Faculty, Hatay, Turkey (Türkiye)

REFERENCES:
- [Result] Sinatra RS, Jahr JS, Reynolds LW, Viscusi ER, Groudine SB, Payen-Champenois C. Efficacy and safety of single and repeated administration of 1 gram intravenous acetaminophen injection (paracetamol) for pain management after major orthopedic surgery. Anesthesiology. 2005 Apr;102(4):822-31. doi: 10.1097/00000542-200504000-00019. PMID 15791113